CLINICAL TRIAL: NCT06172608
Title: Effect of Educational Program on Parental Stress of Parents of Children With Congenital Heart Disease Undergoing Cardiac Surgery: Quasi Experimental Study
Brief Title: Effect of Educational Program on Parental Stress of Parents of Children With CHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, HAMAYUN KHAN, Principal Investigator, Zhengzhou University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023-296
Record Dates: First submitted 2023-11-29; First posted 2023-12-15 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Congenital Heart Defect
Keywords: Congenital Heart disease, parental stress
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (I) (Experimental): Intervention group (I) will be receiving a psychoeducational intervention along with routine care they are getting in the hospital
  Interventions: Other: psychoeducational intervention
- Control group (C) (No Intervention): Comparison usual care and Leaflet of the information. At the end of the trial these also get the video and educational sessions as intervention group.

INTERVENTIONS:
Other: psychoeducational intervention — . Intervention group (I) will receive psychosocial education which will be consist of two parts. 1) Face to Face 2) Community based intervention.
  1. Face to face: This face to face session will be consisting of 30-minute session soon after inclusion into the study. A leaflet consisting of all information will be provided to all the patents taking part in the study.
  2. Community Based Intervention: In community based interventions prerecorded videos about all the topics covered in face to face session will be made available to parents via a secure online platform. Parents can easily browse it easily when they need it. These videos will be recorded in local language (Urdu), which is easy to understand for almost all the people.
  Arms: Intervention Group (I)

SUMMARY:
Congenital Heart disease accounts for about one third of the all congenital anomalies. In last decades' huge advancements occurred in treatment and diagnosis. More and more surgeries are being done which causes stress in parents and affects their mental health. Some studies have reported that about one third of the parents of children with CHD remain in stress even after surgery is being done. The goal of this trial is to evaluate effect of educational intervention on mental health of parents of children with congenital heart disease undergoing cardiac surgery compared to the parents who get usual care and pamphlets of the same information.

The investigators are including parents of children with CHD who are already diagnosed with CHD and are undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of children with congenital heart disease
2. Patient is scheduled for elective cardiac surgery and not had any surgery before.
3. Willing to participate in the study

Exclusion Criteria:

1. Parents of CHD who have other critical conditions along with CHD
2. Parents able to understand local languages (Urdu and Pashto)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Parental stress in parents of children with congenital Heart disease | [Time Frame: INTERVENTION group (I) Baseline (beginning of the study); at 1 day of discharge time and 12 weeks after discharge from hospital].
  Stress changes will be measured via Parental Stress Scale (PSS). The PSS is scored by summing the scores for all 18 items. The total score can range from 18 to 90, with higher scores indicating higher levels of parental stress. The PSS also has two subscales: Child Demandingness (CD) and Parental Competence (PC). PSS scores are interpreted based on the following ranges: 18-37 low stress, 38-56 Moderate stress and 57-90 as high stress.

SECONDARY OUTCOMES:
Changes on parental QoL | [ Time Frame: INTERVENTION group - Baseline (beginning of the study); at 1 day of time of discharge and 12 weeks after intervention. CONTROL group - baseline; at time of discharge and 12 weeks after intervention.]
  Changes on parental quality of life will be assessed through World Health Organization Quality of Life-Bref (WHOQOL-Bref). The WHOQOL-Bref instrument is composed by 26 items, which are organized in 4 specific domains: Physical (7 items), Psychological (6 items), Social Relationships (3 items), Environment (8 items) and a general QoL facet (2 items). All items are quoted from 1 to 5. Three items, related to questions posed negatively (Q3, Q4 and Q26), must be reversed (the calculation implies the subtraction of their value to six units). The results are transformed on a scale of 0 to 100. Each domain score is computed through the formula: [(sum of all items - number of items) / (4x number of items)] x 100. Higher scores correspond to better quality of life.

OTHER OUTCOMES:
Depression in parents of children with CHD | [Time Frame: INTERVENTION group (I) Baseline (beginning of the study); at 1 day of discharge time and 12 weeks after discharge from hospital]
  Depression in parents of children with CHD will be assessed through DASS. The Depression Anxiety Stress Scales (DASS) is a self-report questionnaire that assesses the three most common negative emotional states: depression, anxiety, and stress. It is a widely used tool in research and clinical settings to measure these symptoms and their impact on an individual's well-being. Each item on the DASS is rated on a 4-point Likert scale, ranging from 0 (never) to 3 (almost always). The total score for each subscale is calculated by summing the scores for the items on that subscale. Higher scores on each subscale indicate more severe symptoms.
Anxiety in parents of children with CHD | [Time Frame: INTERVENTION group (I) Baseline (beginning of the study); at 1 day of discharge time and 12 weeks after discharge from hospital]
  Anxiety in parents of children with CHD will be assessed through DASS. The Depression Anxiety Stress Scales (DASS) is a self-report questionnaire that assesses the three most common negative emotional states: depression, anxiety, and stress. It is a widely used tool in research and clinical settings to measure these symptoms and their impact on an individual's well-being. Each item on the DASS is rated on a 4-point Likert scale, ranging from 0 (never) to 3 (almost always). The total score for each subscale is calculated by summing the scores for the items on that subscale. Higher scores on each subscale indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhengzhou University,, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No